CLINICAL TRIAL: NCT02267265
Title: A Randomized Controlled Trial Pilot Study of the Thirty Million Words® Newborn Initiative Intervention, a Novel Postpartum Educational Video
Brief Title: Pilot Study of Novel Postpartum Educational Video Intervention
Acronym: TMW-NI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Opinion Research Center (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TMW-NI
Record Dates: First submitted 2014-09-11; First posted 2014-10-17 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Behavior; Communication; Language
Keywords: educational intervention; language development; universal newborn hearing screening; postpartum; parental attachment; loss to follow-up; hearing loss; achievement gap; language gap; school readiness
MeSH Terms: conditions — Behavior; Communication; Language; Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment intervention (Experimental): The treatment group will complete a demographics questionnaire and the knowledge survey before the intervention. Participants will then view the 10 minute TMW-Newborn Intervention video around the time of the newborn hearing screening. Participants whose newborn does not pass the hearing screen will view an additional 3 minute video detailing the importance of following up for an outpatient re-screening. The participant will complete the knowledge survey again before discharge, and after approximately four to six weeks.
  Interventions: Other: TMW-Newborn Intervention video
- Control intervention (Active Comparator): The control group will complete a demographics questionnaire and knowledge survey. Participants will subsequently view the 10-minute Safe Sleep for your Baby (SIDS) educational video. It is an educational video developed by the National Institute of Child Health and Development (NICHD) promoting the prevention of Sudden Infant Death Syndrome. This will be around the time of the newborn hearing screening. Participants will complete the knowledge survey again before discharge, and after approximately four to six weeks.
  Interventions: Other: Safe Sleep for your Baby (SIDS) educational video

INTERVENTIONS:
Other: TMW-Newborn Intervention video — This is an educational video intervention developed by the Thirty Million Words® Initiative Lab.
  Arms: Treatment intervention
Other: Safe Sleep for your Baby (SIDS) educational video — It is an educational video developed by the National Institute of Child Health and Development (NICHD) promoting the prevention of Sudden Infant Death Syndrome.
  Arms: Control intervention

SUMMARY:
A child's early language environment is pivotal for language development. Disparities in early language environments contribute to the gap in school readiness between poor and more advantaged children. Ultimately this leads to disparities in students' school achievement and economic outcomes. While recent research has highlighted the value of early intervention for children in disadvantaged families, most existing interventions begin too late, reach only a small proportion of children at risk, and do not capitalize on the critical role that parent language plays in a child's educational trajectory. To address this challenge, the investigators propose to develop and evaluate a novel language-based, perinatal public health intervention, Thirty Million Words Newborn Initiative (TMW-NI). It is proposed that new mothers will receive this educational intervention while their babies are undergoing the universal newborn hearing screen. The intervention will use video, animation, and interactive questions to convey the importance of the early language environment and to illustrate strategies parents can use to promote language learning. The investigators will conduct formative research with mothers of low socioeconomic status (low-SES) and with healthcare providers to inform the content and format of the intervention prototype. Also critical for acceptability, the investigators will use an iterative approach to develop the intervention, with review of the work-in-progress by the intended audience. To assess feasibility and initial efficacy, the investigators will conduct a randomized-controlled trial with low-SES mothers during the newborn period. The investigators hypothesize that TMW-NI will positively impact parents' knowledge and beliefs about the role of language input for a child's language development.

ELIGIBILITY:
Inclusion Criteria:

-Postpartum mothers admitted to the mother-baby unit.

Exclusion Criteria:

* Mothers of infants who were admitted to the neonatal intensive care unit (NICU).
* Mothers who experienced any serious medical complications during birth.
* Mothers who do not expect to reside in Illinois for the duration of the study (approximately two months).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in TMW-NI knowledge survey | About 24 hours post intervention
  Scores on the TMW-NI knowledge will be compared to pre-intervention scores.
Change in TMW-NI knowledge survey | About 4 weeks post intervention
  Scores on the TMW-NI knowledge will be compared to pre-intervention scores.

SECONDARY OUTCOMES:
Loss to follow-up | About 4 weeks post intervention
  Measuring change in loss to follow-up statistics for patients that do not pass the universal newborn hearing screening.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, MD, Principal Investigator — The University of Chicago Medicine; Kristin Leffel, AB, Study Chair — The University of Chicago Medicine
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois

REFERENCES:
- [Derived] Sowa LE, Thomas JMN, Hundertmark AC, Baroody FM, Suskind DL. Leveraging the universal newborn hearing screen to impact parental knowledge of childhood speech development in low socioeconomic populations: A randomized clinical trial. Int J Pediatr Otorhinolaryngol. 2021 Jul;146:110763. doi: 10.1016/j.ijporl.2021.110763. Epub 2021 May 11. PMID 34000494